CLINICAL TRIAL: NCT00700570
Title: An Open Label Study to Assess the Resection Rate of Liver Metastases Following Neoadjuvant Therapy With Avastin in Combination With Oxaliplatin and Capecitabine (XELOX) in Patients With Metastatic Colorectal Cancer With Unresectable Liver Metastasis
Brief Title: A Study of Avastin (Bevacizumab) in Combination With XELOX in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21209
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: oxaliplatin

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5mg/kg iv on day 1 of each 2 week cycle.
Drug: capecitabine [Xeloda] — 1000mg/m2 iv on days 1-5 and 8-12 of each 2 week cycle
Drug: oxaliplatin — 85mg/m2 iv on day 1 of each 2 week cycle

SUMMARY:
This single arm study will assess the resection rate of liver metastasis, time to disease progression, and safety of neoadjuvant treatment with Avastin in combination with oxaliplatin and capecitabine (XELOX) in patients with metastatic colorectal cancer with unresectable liver metastasis. Patients will receive Avastin 5mg/kg iv on day 1 of every 2 week cycle, oxaliplatin 85mg/m2 iv on day 1 of every 2 week cycle, and capecitabine 1000mg/m2 on days 1-5 and 8-12 of every 2 week cycle. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, <=75 years of age;
* chemotherapy-naive for stage IV colorectal cancer with unresectable liver metastasis;
* >=1 measurable lesion;
* ECOG status 0-2.

Exclusion Criteria:

* prior exposure to Avastin;
* clinical or radiological evidence of CNS metastases;
* uncontrolled hypertension, or clinically significant cardiovascular disease;
* ongoing treatment with aspirin (>325mg/day) or other medications known to predispose to gastrointestinal ulceration.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Taiwan (4):
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan

RESULTS

PARTICIPANT FLOW:
Groups:
- Resected: Participants with unresectable liver metastases secondary to colorectal cancer (CRC) were assigned to receive neoadjuvant treatment of intravenous (IV) bevacizumab with oral (PO) capecitabine and IV oxaliplatin (XELOX). Bevacizumab was given as 5 milligrams per kilogram (mg/kg) on Day 1 of each 14-day cycle during Cycles 1 to 5 and/or Cycles 8 to 12. During Cycles 1 to 12, IV oxaliplatin was given as 85 milligrams per meter-squared (mg/m^2) on Day 1, and PO capecitabine as 1000 mg/m^2 twice daily on Days 1 to 5 and 8 to 12. Resectability was assessed at completion of Cycle 5. Resectable participants followed a new algorithm: complete Cycle 6 (XELOX), rest for 4 weeks, undergo surgery, rest for 4 weeks, complete adjuvant therapy during Cycles 7 (XELOX) and 8 to 12 (bevacizumab plus XELOX), and continue an additional 6 cycles with capecitabine and bevacizumab per Investigator discretion. Participants could be withdrawn at any point for unacceptable toxicity.
- Unresected: Participants with unresectable liver metastases secondary to CRC were assigned to receive neoadjuvant treatment of IV bevacizumab with XELOX. Bevacizumab was given as 5 mg/kg on Day 1 of each 14-day cycle during Cycles 1 to 5 and/or Cycles 8 to 12. During Cycles 1 to 12, IV oxaliplatin was given as 85 mg/m^2 on Day 1, and PO capecitabine as 1000 mg/m^2 twice daily on Days 1 to 5 and 8 to 12. Resectability was assessed at completion of Cycle 5. Unresectable participants with partial response (PR) or stable disease (SD), according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, repeated neoadjuvant treatment until documented resectability or progressive disease (PD). Participants could be withdrawn at any point for unacceptable toxicity.
Period: Overall Study
Arm/Group | Resected | Unresected
Started | 19 | 26
Completed | 8 | 0
Not Completed | 11 | 26
Not completed — Adverse Event | 2 | 6
Not completed — Discretion of Investigator or Sponsor | 0 | 3
Not completed — Disease Progression | 8 | 11
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Resected: Participants with unresectable liver metastases secondary to CRC were assigned to receive neoadjuvant treatment of IV bevacizumab with XELOX. Bevacizumab was given as 5 mg/kg on Day 1 of each 14-day cycle during Cycles 1 to 5 and/or Cycles 8 to 12. During Cycles 1 to 12, IV oxaliplatin was given as 85 mg/m^2 on Day 1, and PO capecitabine as 1000 mg/m^2 twice daily on Days 1 to 5 and 8 to 12. Resectability was assessed at completion of Cycle 5. Resectable participants followed a new algorithm: complete Cycle 6 (XELOX), rest for 4 weeks, undergo surgery, rest for 4 weeks, complete adjuvant therapy during Cycles 7 (XELOX) and 8 to 12 (bevacizumab plus XELOX), and continue an additional 6 cycles with capecitabine and bevacizumab per Investigator discretion. Participants could be withdrawn at any point for unacceptable toxicity.
- Unresected: Participants with unresectable liver metastases secondary to CRC were assigned to receive neoadjuvant treatment of IV bevacizumab with XELOX. Bevacizumab was given as 5 mg/kg on Day 1 of each 14-day cycle during Cycles 1 to 5 and/or Cycles 8 to 12. During Cycles 1 to 12, IV oxaliplatin was given as 85 mg/m^2 on Day 1, and PO capecitabine as 1000 mg/m^2 twice daily on Days 1 to 5 and 8 to 12. Resectability was assessed at completion of Cycle 5. Unresectable participants with PR or SD, according to RECIST version 1.1, repeated neoadjuvant treatment until documented resectability or PD. Participants could be withdrawn at any point for unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Resected | Unresected | Total
Number analyzed (Participants) | 19 | 26 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.6) | 55.1 (10.4) | 55.08 (11.2)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Conversion From Unresectable to Resectable Liver Metastases
Description: Participants were assessed via microscopic and macroscopic examination for tumor resectability after completion of 5 cycles of neoadjuvant treatment. Unresectable participants exhibited any of the following criteria: greater than or equal to (≥) 4 liver metastases; location and/or distribution of metastatic disease within the liver considered unsuitable for resection with clear margins; liver involvement precluding resection, in the setting of adequate parenchymal volume for otherwise viable liver function in the immediate postoperative period; and inability to maintain adequate circulation for viable liver function. Participants who had not met any of the above criteria at the end of 5 cycles underwent surgical resection. The percentage of participants with conversion from initially unresectable to resectable liver metastases was calculated as [number of participants eligible for surgical resection divided by the number analyzed] multiplied by 100.
Time Frame: After 5 cycles of neoadjuvant treatment (10 weeks)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Participants with unresectable liver metastases secondary to CRC were assigned to receive neoadjuvant treatment of IV bevacizumab with XELOX. Bevacizumab was given as 5 mg/kg on Day 1 of each 14-day cycle during Cycles 1 to 5 and/or Cycles 8 to 12. During Cycles 1 to 12, IV oxaliplatin was given as 85 mg/m^2 on Day 1, and PO capecitabine as 1000 mg/m^2 twice daily on Days 1 to 5 and 8 to 12. Resectability was assessed at completion of Cycle 5. Resectable participants followed a new algorithm: complete Cycle 6 (XELOX), rest for 4 weeks, undergo surgery, rest for 4 weeks, complete adjuvant therapy during Cycles 7 (XELOX) and 8 to 12 (bevacizumab plus XELOX), and continue an additional 6 cycles with capecitabine and bevacizumab per Investigator discretion. Unresectable participants with PR or SD, according to RECIST version 1.1, repeated neoadjuvant treatment until documented resectability or PD. Participants could be withdrawn at any point for unacceptable toxicity.
Arm/Group | All Participants
Number analyzed (Participants) | 45
percentage of participants | 42.2

2. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Objective tumor response was assessed using RECIST version 1.1. Disease progression was defined as a ≥20 percent (%) increase in the sum of longest diameters of target lesions, taking as reference the smallest sum obtained at previous tumor assessment, or the appearance of any new lesions. The percentage of participants with disease progression was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 3 years (at Baseline, end of Cycle 5, time of surgery, and within 4 weeks of end of treatment [EOT])
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Resected | Unresected
Number analyzed (Participants) | 19 | 26
percentage of participants | 52.6 | 46.2

3. Secondary Outcome: Time to Disease Progression
Description: Objective tumor response was assessed using RECIST version 1.1. Disease progression was defined as a ≥20% increase in the sum of longest diameters of target lesions, taking as reference the smallest sum obtained at previous tumor assessment, or the appearance of any new lesions. Time to disease progression was defined as the time from first dose to time of disease progression. Participants without progression were censored at the time of last tumor assessment. Time to disease progression was estimated using Kaplan-Meier analysis and expressed in months.
Time Frame: Up to approximately 3 years (at Baseline, end of Cycle 5, time of surgery, and within 4 weeks of EOT)
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Resected | Unresected
Number analyzed (Participants) | 19 | 26
months | 10.1 [7.0 to 20.4] | 8.7 [5.0 to 14.2]
Statistical Analysis 1: Comparison: Resected vs Unresected; Test type: Superiority or Other; p = 0.1341, Log Rank

4. Secondary Outcome: Percentage of Participants With a Best Overall Tumor Response of Complete Response (CR) or PR According to RECIST Version 1.1
Description: Objective tumor response was assessed using RECIST version 1.1. CR was defined as the disappearance of all target lesions, and PR was defined as a ≥30% decrease in the sum of longest diameters compared to Baseline. Response was confirmed at a minimum of 4 weeks after the first documented response. The percentage of participants with confirmed CR or PR was calculated as [number of participants meeting the respective criteria divided by the number analyzed] multiplied by 100.
Time Frame: Up to approximately 3 years (at Baseline, end of Cycle 5, time of surgery, within 4 weeks of EOT, and at least 4 weeks after initial response)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Resected | Unresected
Number analyzed (Participants) | 19 | 26
percentage of participants | 47.4 | 34.6

5. Secondary Outcome: Percentage of Participants by Best Overall Tumor Response According to RECIST Version 1.1
Description: Objective tumor response was assessed using RECIST version 1.1. CR was defined as the disappearance of all target lesions, and PR was defined as a ≥30% decrease in the sum of longest diameters compared to Baseline. Response was to be confirmed at a minimum of 4 weeks after the first documented response. Stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, as well as no new target lesions. Disease progression or PD was defined as a ≥20% increase in the sum of longest diameters of target lesions, taking as reference the smallest sum obtained at previous tumor assessment, or the appearance of any new lesions. Non-evaluability for tumor assessment was also documented when applicable. The percentage of participants with each level of response was calculated as [number of participants meeting the respective criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 4
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Resected | Unresected
Number analyzed (Participants) | 19 | 26
percentage of participants
  CR | 36.8 | 0
  PR | 10.5 | 34.6
  SD | 0 | 15.4
  PD | 52.6 | 46.2
  Non-evaluable | 0 | 3.8
Statistical Analysis 1: Comparison: Resected vs Unresected; Test type: Superiority or Other; p = 0.0010, Fisher Exact

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years (continuously until 4 weeks after EOT)
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=45)
Diarrhoea (Gastrointestinal disorders) | 3
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 2
Enterocolitis infectious (Infections and infestations) | 1
Perihepatic abscess (Infections and infestations) | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=45)
Anaemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 17
Fatigue (General disorders) | 18
Mucosal inflammation (General disorders) | 8
Pyrexia (General disorders) | 8
Paronychia (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 20
Dizziness (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 19
Peripheral sensory neuropathy (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 9
Proteinuria (Renal and urinary disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 35
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.